CLINICAL TRIAL: NCT01953289
Title: Importance of Peritoneal Free Fluid Cultures in Both Perforated and Non-perforated Appendicitis
Brief Title: Importance of Peritoneal Free Fluid Cultures in Acute Appendicitis
Acronym: IFFSA
Status: Withdrawn | Type: Observational
Why Stopped: Sub investigator is working no longer in the hospital. No participants were enrolled.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S-54473
Record Dates: First submitted 2013-02-19; First posted 2013-09-30 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Appendicitis
Keywords: Appendicitis; Free fluid
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Appendicitis: Free fluid in perforated or non-perforated appendicitis

SUMMARY:
The purpose of this study is to evaluate the frequency of positive free fluid cultures in both perforated and non-perforated appendicitis. In addition predictors of positive free fluid cultures will be analyzed.

DETAILED DESCRIPTION:
Prior to surgery, all patients will receive antibioprophylaxis. In case of free peritoneal fluid, a sample is aspirated and sent for microbiology. A lavage with saline is not necessary. The decision to start postoperative antibiotic is left at the discretion of the surgeon. The decision to leave an abdominal drain is left at the discretion of the surgeon.

The use of a preoperative single dose administration of antibiotics has been extensively studied and found beneficial in the prevention of SSI in appendicitis. However, the use of continued postoperative antibiotics has barely been studied. The sparse evidence that exist does not seem to support its systematic use. During appendectomy the surgeon frequently encounters turbid free fluid, even in non-perforated appendicitis. It is common practice in Belgium to continue antibiotic prophylaxis for 5 days after aspiration and lavage. Although the aspect often seems purulent, it is unknown in what percentage this fluid is contaminated. Also, it is unknown whether after aspiration and lavage intra-abdominal drains are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Appendicitis (Perforated/ Non-perforated) Free fluid Age: 6 - 90y

Exclusion Criteria:

* Immunosuppression (recent chemotherapy, chronic use of immunosuppressive medication) Age < 6 and > 90y

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with perforated or non-perforated appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the frequency of positive free fluid cultures in both perforated and non-perforated appendicitis | 24 hours
  In case of free peritoneal fluid, a sample will be aspirated and sent for microbiology.

CONTACTS AND LOCATIONS:
Overall Officials: André JL D'Hoore, PhD, Principal Investigator — university Clinics Gasthuisberg department of abdominal surgery
Locations (1):
- University Clinics Gasthuisberg, Leuven, Flemish Brabant, Belgium